CLINICAL TRIAL: NCT05630105
Title: National Cohort of Patients With Cowden's Disease and With a Constitutional Alteration of the PTEN Gene for the Prospective Assessment of the Risk of Cancer.
Brief Title: Cancer Risk Assessment in Patients With a Constitutional Alteration of the PTEN Gene
Acronym: COCO
Status: Recruiting | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB2022-02
Record Dates: First submitted 2022-11-10; First posted 2022-11-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: PTEN Gene Mutation
Keywords: PTEN gene mutation; risk of cancer occurence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicentric, observational, retrospective and prospective study, aiming to estimate the risk of cancer occurrence in subjects carrying a PTEN mutation, based on the constitution of a national cohort.

DETAILED DESCRIPTION:
After collection of the non objection and verification of the eligibility criteria, a first clinical questionnaire will be completed by the participant and the prescribing physician to collect the main medical events including the history of malignant tumor pathologies until the date of inclusion in the study.

Thereafter, an annual questionnaire will be sent to the participants to update the elements related to a tumor pathology.

For the case of patients who have died or been lost to follow-up, only the information from the first clinical questionnaire will be collected from the data available from the prescribing physician without informing the relatives. However, the investigating center will have to check that these patients have not objected, during their lifetime, to the use of their data.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Adult or child without age limit.
3. Carrier of a constitutional or mosaic alteration of the PTEN gene established and/or confirmed by the Institut Bergonié's genetics laboratory, following a request for molecular diagnosis made between 1997 and 2027.
4. Participant informed of his genetic diagnosis.
5. Participant informed and not having expressed non-opposition to participate in the research.
6. Participant affiliated to a French social security system in accordance with French law on research involving the human person.

Exclusion Criteria:

1. Participant under guardianship or curatorship. Exception: a participant with autism may be included in the study.
2. Persons deprived of their liberty by a judicial or administrative decision.
3. Persons under psychiatric care, persons admitted to a health or social establishment for purposes other than research; Exception: a participant with autism may be included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: National observational cohort of participants identified as carriers of a constitutional alteration of the PTEN gene identified and/or confirmed by the Bergonié Institute, the national reference laboratory for the molecular diagnosis of Cowden's disease between 1997 and 2027.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2048-01 (Estimated); Study Completion 2048-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with a cancer event | From date of identification of a constitutional alteration of the PTEN gene until the date of first cancer event or date of death from any cause, whichever came first, assessed up to 20 years.
  Number of subjects with a cancer event (any cancer) observed in the population of subjects presenting a constitutional alteration of the PTEN gene.

SECONDARY OUTCOMES:
Number of subjects with a breast cancer event | From date of identification of a constitutional alteration of the PTEN gene until the date of first breast cancer event or date of death from any cause, whichever came first, assessed up to 20 years.
  Number of subjects with a breast cancer event (any cancer) observed in the population of subjects presenting a constitutional alteration of the PTEN gene.
Number of subjects with a thyroid cancer event | From date of identification of a constitutional alteration of the PTEN gene until the date of first thyroid cancer event or date of death from any cause, whichever came first, assessed up to 20 years.
  Number of subjects with a thyroid cancer event (any cancer) observed in the population of subjects presenting a constitutional alteration of the PTEN gene.
Number of subjects with an endometrial cancer event | From date of identification of a constitutional alteration of the PTEN gene until the date of first endometrial cancer event or date of death from any cause, whichever came first, assessed up to 20 years.
  Number of subjects with an endometrial cancer event (any cancer) observed in the population of subjects presenting a constitutional alteration of the PTEN gene.
Number of subjects with a renal cancer event | From date of identification of a constitutional alteration of the PTEN gene until the date of first renal cancer event or date of death from any cause, whichever came first, assessed up to 20 years.
  Number of subjects with a renal cancer event (any cancer) observed in the population of subjects presenting a constitutional alteration of the PTEN gene.
Number of subjects with a colorectal cancer event | From date of identification of a constitutional alteration of the PTEN gene until the date of first colorectal cancer event or date of death from any cause, whichever came first, assessed up to 20 years.
  Number of subjects with a colorectal cancer event (any cancer) observed in the population of subjects presenting a constitutional alteration of the PTEN gene.
Number of subjects with a melanoma cancer event | From date of identification of a constitutional alteration of the PTEN gene until the date of first melanoma cancer event or date of death from any cause, whichever came first, assessed up to 20 years.
  Number of subjects with a melanoma cancer event (any cancer) observed in the population of subjects presenting a constitutional alteration of the PTEN gene.

CONTACTS AND LOCATIONS:
Overall Officials: Virginie BUBIEN, Dr, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Comprehensive Cancer Center, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No